CLINICAL TRIAL: NCT06184633
Title: DUTCH Weight Control in Atrial Fibrillation Study, a Multi-center, Double-blind, Randomized, Parallel Group, Placebo-controlled Trial
Brief Title: DUTCH Weight Control in Atrial Fibrillation Study
Acronym: DUTCH-WAIST
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Ron Pisters, Head of Cardioresearch and principal investigator, dr. R. Pisters, Rijnstate Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U1111-1275-9989
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Atrial Fibrillation; Obesity; Weight Loss
MeSH Terms: conditions — Atrial Fibrillation; Obesity; Weight Loss | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Semaglutide injections + combined lifestyle intervention
  Interventions: Drug: Semaglutide 3.2 MG/ML
- Placebo (Placebo Comparator): Placebo Semaglutide injections + combined lifestyle intervention
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide 3.2 MG/ML — Intervention arm receives semaglutide in addition to combined lifestyle intervention
  Arms: Intervention
Drug: Placebo — Control arm receives placebo in addition to combined lifestyle intervention
  Arms: Placebo

SUMMARY:
Quantify the effect of an innovative weight loss management on rhythm control.

DETAILED DESCRIPTION:
Rationale: Weight reduction promotes reversed atrial remodeling in obese AF patients.

Objective: Quantify the effect of an innovative weight loss management on rhythm control.

Study design: Multi-center, double-blind, randomized, parallel group, placebo-controlled trial of semaglutide 2.4 mg versus placebo.

Study population: Adults with obesity and new onset persistent AF scheduled for electrical cardioversion.

Intervention: semaglutide 2.4 mg subcutaneous (s.c.) once weekly (index) compared to placebo (control), at the background of standard obesity treatment (combined lifestyle intervention) and cardiology follow-up management in both arms.

Main study parameters/endpoints: The primary efficacy clinical endpoint of the trial is assessed at 12 months by a 7 point scale. Only the worst clinical outcome will be retained as the primary efficacy outcome. The 7 mutually exclusive outcomes hierarchically ranked from worst to best are:

* Arrhythmic death while using anti-arrhythmic drugs (Vaughn-Williams class I or III)*
* AF despite pulmonary vein isolation
* AF despite current use of anti-arrhythmic drugs (Vaughn-Williams class I or III)
* AF without a pulmonary vein isolation and without the current use of anti-arrhythmic drugs (Vaughn-Williams class I or III)
* Sinus rhythm on the 12-lead ECG with the use of a pulmonary vein isolation
* Sinus rhythm on the 12-lead ECG with current use of anti-arrhythmic drugs (Vaughn-Williams class I or III)
* Sinus rhythm on the 12-lead ECG without the current use of anti-arrhythmic drugs (Vaughn-Williams class I or III) and without a pulmonary vein isolation

  * When LTFU or death other than anti-arrhythmic death, last known rhythm will be used.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic, first detected (at maximum 6 months prior to enrollment) persistent AF -
* Age ≥ 18
* Obesity, as defined as:

  * BMI ≥ 30 kg/m2, or
  * BMI ≥27 kg/m2 with the presence of at least one weight related comorbidity (treated or untreated, e.g. hypertension, dyslipidaemia, obstructive sleep apnea, cardiovascular disease)
* Scheduled ECV
* Written informed consent

Exclusion Criteria:

* Permanent AF
* Secondary AF, i.e. due to thyrotoxicosis, infection (e.g. pneumonia) or post-(cardiothoracic) surgery
* Current or previous treatment with amiodaron
* HbA1c ≥ 48 mmol/L, <3 months prior to randomization
* History of diabetes mellitus type 1 or 2
* Prior bariatric surgery
* Use of other anti-obesity medication, <3 months prior to enrollment
* Contra-indication for, or prior use of a GLP1-receptor agonist
* History of chronic pancreatitis or acute pancreatitis <6 months
* Acute coronary syndrome <6 months
* Severe (grade III) valvular disease
* eGFR <30 mL/min/1.73m2
* Heart failure NYHA class III-IV
* Participation in another investigational drug or device study in the past 30 days (registry enrollment is allowed)
* Any condition or therapy, which would make the participant unsuitable for the study (e.g. vulnerable, non-compliance) or life-expectancy <12 months, as judged by the treating physician.
* Female who is pregnant, breastfeeding, intends to become pregnant, or is of child-bearing potential and not using a highly effective contraceptive method.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-07-21 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy clinical endpoint of the trial is assessed at 12 months by a 7 point scale. Only the worst clinical outcome will be retained as the primary efficacy outcome | At 1 year follow-up
  The 7 mutually exclusive outcomes hierarchically ranked from worst to best are:
  * Arrhythmic death while using anti-arrhythmic drugs (Vaughn-Williams class I or III)*
  * AF despite pulmonary vein isolation
  * AF despite current use of anti-arrhythmic drugs (Vaughn-Williams class I or III)
  * AF without a pulmonary vein isolation and without the current use of anti-arrhythmic drugs (Vaughn-Williams class I or III)
  * Sinus rhythm on the 12-lead ECG with the use of a pulmonary vein isolation
  * Sinus rhythm on the 12-lead ECG with current use of anti-arrhythmic drugs (Vaughn-Williams class I or III)
  * Sinus rhythm on the 12-lead ECG without the current use of anti-arrhythmic drugs (Vaughn-Williams class I or III) and without a pulmonary vein isolation
    * When LTFU or death other than anti-arrhythmic death, last known rhythm will be used.

SECONDARY OUTCOMES:
Change in AF related symptoms measured by the modified EHRA classification between the index visit and at 12 months after the index visit. | week 0 and 52
  EHRA: European Heart Rythm Association
  1= no symptoms 2a= mild symptoms; Normal dialy activity not affected, symptoms not troublesome to patient 2b= moderate symptoms; Normal daily activity not affected but patient troubled by symptoms 3= severe symptoms; Normal daily activity affected 4= disabling symptoms; Normal daily activity discontinued
Change in quality of life measured by the EQ-5D-5L between the index visit and at 12 months after the index visit. | week 0 and 52
  Descriptive system for health-related quality of life states in adults, consisting of five dimensions (Mobility, Self-care, Usual activities, Pain & discomfort, Anxiety & depression), each of which has five severity levels that are described by statements appropriate to that dimension.
  LEVEL 1: indicating no problem LEVEL 2: indicating slight problems LEVEL 3: indicating moderate problems LEVEL 4: indicating severe problems LEVEL 5: indicating unable to/extreme problems
Number of hospitalizations because of an AF recurrence. | week 0-52
Number of unscheduled hospital visits because of adverse events of AAD. | week 0-52
Number of scheduled electrical cardioversions. | week 0-52
Number of unscheduled electrical cardioversions. | week 0-52
Number of intravenous chemical cardioversions (using Vaughan-Williams class I drugs). | week 0-52
Total number of unscheduled cardioverions. | week 0-52
Change in waist circumference, measured in cm | week 0 and 52
Change in weight, measured in % and kg | week 0 and 52
Change in BMI, measured in kg/m2 | week 0 and 52

CONTACTS AND LOCATIONS:
Overall Officials: Ron Pisters, dr., Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No